CLINICAL TRIAL: NCT02955056
Title: A Feasibility Study to Explore the Difference in Healing Time Between Teriparatide Treatment and Standard Care on Weber B Ankle Fractures in Older People
Brief Title: Ankle Fractures Treated With Teriparatide
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13OR006; 2015-005423-32 (EudraCT Number); 143755 (Other: IRAS)
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Fracture, Ankle
Keywords: Weber B
MeSH Terms: conditions — Ankle Fractures | interventions — Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teriparatide Intervention (Experimental): Will be asked to self-administer Teriparatide treatment (self-injection) once a day for 12 weeks
  Interventions: Drug: Forsteo
- Usual care (No Intervention): No intervention, patients will be treated as per local practice but will be followed up identically to the intervention group.

INTERVENTIONS:
Drug: Forsteo — 20 micrograms/80 microlitres solution for injection in pre-filled pen
  Other Names: Teriparatide hormone
  Arms: Teriparatide Intervention

SUMMARY:
This is a single site feasibility trial to test whether daily administration of Teriparatide, in participants with Weber type B ankle fractures that are being conservatively managed, is superior to the standard care treatment with regard to the rate of healing.

DETAILED DESCRIPTION:
Ankle fractures are common in older people, they are very disabling and require either a cast or a boot for treatment and the patients need to use crutches for balance. These fractures can lead to complications including non union or delayed union in addition to risks of clotting of the leg vessels (deep vein thrombosis) where these clots can dislodge and migrate to the lungs (pulmonary embolus) resulting in breathing difficulties and/or death. Also these fractures commonly result in patients needing a temporary period of residential care. Therefore, if the healing time can be reduced, there is a potential for large benefits for the patient and reduced care costs for health and social care services.

Teriparatide hormone is one of the new medications used for treating osteoporosis(weak bones), and studies in the USA have reported that Teriparatide hormone treatment can accelerate bone fracture healing time in pelvic fractures.

Other reports also support faster healing time when Teriparatide hormone is used.

The investigators are carrying out this feasibility study with 10 participants, in order to provide the information that will prepare us for carrying out a definitive study in the future.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female (women of non-child bearing potential only*), aged 50 years or above
* Ankle fracture Weber type B suitable for conservative treatment in a synthetic cast
* The fracture should be less than 10 days old
* Blood test results within the normal range as defined by Nottingham University Hospitals NHS Trust (FBC, ESR, LFT, RFT, PTH, Bone profile (Calcium, albumin, total protein and alkaline phosphatase) and thyroid function)
* Able and willing to comply with all study requirements

Exclusion Criteria:

* Current smokers (both tobacco and electronic cigarettes)
* Chronic renal disease
* Insulin dependent diabetes mellitus
* History of hypercalcemia
* End stage liver disease (liver cirrhosis)
* Patient with any current or past history of cancer
* Use of bisphosphonates, Zolendronic acid or fluorides within the last 6 months
* Any bone conditions other than osteoporosis
* Unable to get out of a chair or bed and walk without the help of another person pre ankle fracture (walking aids are acceptable)
* Contraindication to Teriparatide hormone:
* Hypersensitivity
* High risk of Osteosarcoma, (Paget's disease, chondromas, exposure to radiation, unexplained alkaline phosphatase, etc.)
* Female participants of child-bearing potential, who are pregnant, lactating or planning pregnancy during course of study
* Scheduled elective surgery or other procedures requiring general anaesthesia during the study
* Terminally ill
* Planned blood donor donation during the study
* Participated in another research study involving an investigational product in the past 12 weeks
* Prior external beam of radiation or implant of radiation therapy to the skeleton.
* Any blood diseases leading to a bleeding tendency
* On Heparin, Warfarin or any Anticoagulants

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of healing parameters of the fracture | Week 1 - Week 13
  Assessment of healing parameters of the fracture as identified on the CT scan at Trial Visits

SECONDARY OUTCOMES:
Identify the participant's pain during the treatment period | Week 1 - Week 13
  Pain scores on weight bearing, as assessed by 10-point visual analogue pain score scale
Functional assessment of the ankle using Olerud and Molander questionnaire | Week 7 - Week 13
  measure ankle function at the end of brace/cast treatment

CONTACTS AND LOCATIONS:
Overall Officials: Angus Wallace, Study Chair — Nottingham University Hospitals NHS Trust
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD